CLINICAL TRIAL: NCT05706597
Title: Clinical Relevance of Small Airways Disease in Severe Asthma Patients Treated With Anti-InterLeukin-5 Therapy
Acronym: SAIL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Sponsor
Other Study IDs: SAIL2022
Record Dates: First submitted 2023-01-23; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2022-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this research is to investigate the extent and clinical relevance of small airways disease in severe eosinophilic asthma patients treated with anti-IL5/5R therapy.

ELIGIBILITY:
Inclusion Criteria:

* Severe asthma patients treated with anti-IL5/5R therapy (i.e. mepolizumab, benralizumab, reslizumab) for at least 4 months.

Exclusion Criteria:

* No information about lung function at baseline, or after both 4 months and 12 months.
* No information about clinical response (i.e. number of exacerbations, reduction of mOCS/ maintenance oral corticosteroid dose, ACQ, AQLQ) after both 4 months and 12 months.
* Treatment with another anti-IL5/5R therapy before

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of all severe eosinophilic asthma patients in the MCL, treated with anti-IL5/5R therapy (i.e. mepolizumab, benralizumab, reslizumab) for at least 4 months.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Is change in FEF25-75 during anti-IL5/5R treatment associated with change in asthma control (measured with the asthma control questionnaire -ACQ-) in severe eosinophilic asthma patients after 4 months and after 12 months treatment? | 4 months and 12 months
  Is change in FEF25-75 during anti-IL5/5R treatment associated with change in asthma control (measured with the asthma control questionnaire -ACQ-) in severe eosinophilic asthma patients after 4 months and after 12 months treatment?

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Center Leeuwarden, Leeuwarden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided